CLINICAL TRIAL: NCT01784562
Title: An Open-label Phase IIIb Study of Riociguat in Patients With In-operable CTEPH, or Recurrent or Persisting PH After Surgical Treatment Who Are Not Satisfactorily Treated and Cannot Participate in Any Other CTEPH Trial
Brief Title: Riociguat in Patients With Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Acronym: EAS
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16097; 2012-002104-40 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Chronic thromboembolic pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

INTERVENTIONS:
Drug: Adempas (Riociguat, BAY63-2521) — Individual dosing of riociguat between 0.5 and 2.5 mg three times daily based on patient's well being and blood pressure. (The individual optimal dose should be determined during the initial 8-week titration phase based on patient's monitoring of systolic blood pressure and well-being.)

SUMMARY:
The aim of the study is to assess safety, tolerability and clinical effects of different doses of riociguat in patients with inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH) and who are not satisfactorily treated and cannot participate in any other CTEPH trial. In the US the study runs as an Expanded Access program under 21 CFR 312.320.

ELIGIBILITY:
Inclusion Criteria:

- Male and female patients with CTEPH either inoperable or with persistent or recurrent PH after surgery

Exclusion Criteria:

* All types of pulmonary hypertension other than Dana Point Classification Group 4
* Operable patients listed for PEA (Pulmonary Endarterectomy)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (97):
- United States (23):
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Sacramento, California
  - Aurora, Colorado
  - Weston, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Omaha, Nebraska
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Fairfield, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
- Austria (3):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Vienna, Vienna
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Canada (5):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Colombia (5):
  - Bogotá, Bogota D.C.
  - Bogotá, Cundinamarca
  - Cali, Valle del Cauca Department
  - Bogotá
  - Santa Fé
- Prague, Czechia
- Aarhus N, Denmark
- France (9):
  - Besançon
  - Brest
  - Bron
  - Caen
  - Le Kremlin-Bicêtre
  - Montpellier
  - Pessac
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Hamburg, Hamburg
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
- Italy (3):
  - Pavia
  - Roma
  - Trieste
- Japan (4):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Sendai, Miyagi
  - Bunkyo-ku, Tokyo
- Mexico (3):
  - Mexico City, Mexico City
  - México D.F., Mexico City
  - Monterrey, Nuevo León
- Netherlands (3):
  - Amsterdam
  - Nieuwegein
  - Rotterdam
- Portugal (4):
  - Coimbra, Coimbra District
  - Lisbon, Lisbon District
  - Almada
  - Lisbon
- Russia (2):
  - Novosibirsk
  - Saint Petersburg
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Seville, Sevilla
- Sweden (3):
  - Linköping
  - Lund
  - Umeå
- Switzerland (4):
  - Bern, Canton of Bern
  - Sankt Gallen, Canton of St. Gallen
  - Lausanne, Canton of Vaud
  - Zurich, Canton of Zurich
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (4):
  - Cambridge, Cambridgeshire
  - Sheffield, South Yorkshire
  - Newcastle upon Tyne, Tyne and Wear
  - Glasgow, West Dunbartonshire

REFERENCES:
- [Derived] McLaughlin VV, Jansa P, Nielsen-Kudsk JE, Halank M, Simonneau G, Grunig E, Ulrich S, Rosenkranz S, Gomez Sanchez MA, Pulido T, Pepke-Zaba J, Barbera JA, Hoeper MM, Vachiery JL, Lang I, Carvalho F, Meier C, Mueller K, Nikkho S, D'Armini AM. Riociguat in patients with chronic thromboembolic pulmonary hypertension: results from an early access study. BMC Pulm Med. 2017 Dec 28;17(1):216. doi: 10.1186/s12890-017-0563-7. PMID 29282032